CLINICAL TRIAL: NCT05527665
Title: Sexual Fonction and Discomfort in Women After Midurethral Sling Surgery, Using PPSSQ
Acronym: SEXBSU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0301
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Women over 90 years of age Women who have received a suburethral sling at CHUGA in the gynecology or urology departments between January 2015 and June 2020.
  Women who agreed to complete the PPSSQ
  Interventions: Procedure: Midurethral sling surgery
- Healthy volunteers group: -Adult women under 90 years of age, matched on age and menopausal status to the patient group Women who have never had surgery for stress urinary incontinence with a sub-urethral sling.
  Women who agreed to complete the PPSSQ

INTERVENTIONS:
Procedure: Midurethral sling surgery — This treatment consists of the placement of a sub-urethral sling, usually made of polypropylene, in order to support the urethra during efforts and thus to avoid leaks linked to its hyper mobility. This is a frequent and rapid surgery, which is performed on an outpatient basis. The sling is placed under the patient's urethra with the help of an awl.
  Groups: Patient group

SUMMARY:
Evaluation of the sexual quality of life of women who had a sub-urethral sling several years ago, using a recently validated questionnaire: the PPSSQ (Pelvi-Perineal Surgery Sexuality Questionnaire).

This questionnaire is specifically oriented for women who have undergone surgery for stress urinary incontinence or prolapse. It contains questions specific to post-surgical issues that are not present in other sexual quality of life questionnaires. The questionnaire will also be administered to a group of control women who have not had suburethral sling surgery in order to compare their responses to those of women who have had surgery.

The hypothesis is that the placement of a suburethral sling for stress urinary incontinence increases the quality of sexual life of the women.

ELIGIBILITY:
Inclusion Criteria:

Patient group

* Women who have received a suburethral sling at CHUGA in the gynecology or urology departments between January 2015 and June 2020.
* Women who agreed to complete the PPSSQ

Healthy volunteers group

* Adult women matched on age and menopausal status to the patient group
* Women who have never undergone surgery for stress urinary incontinence by placing a sub-urethral tape.
* Women who agreed to complete the PPSSQ

Exclusion Criteria:

Patient group

* Tape removal.
* Death since surgery.
* Factors that make it impossible to understand the questionnaires: neurological or psychiatric pathology that limits the understanding of the questions, lack of mastery of the French language, illiteracy.
* Absence of perineal sensation.
* Persons referred to in articles L1121-5 to L1121-8 of the CSP.

Healthy volunteers group

* Factors that make it impossible to understand the questionnaires: neurological or psychiatric pathology that limits the understanding of the questions, lack of mastery of the French language, illiteracy.
* Absence of perineal sensation.
* Persons referred to in articles L1121-5 to L1121-8 of the CSP.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have received a sub-urethral sling at CHUGA in the gynecology and urology departments between January 2015 and June 2020.
  Healthy volunteers who agreed to answer the questionnaire fitted on age and menopausal status.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sexual discomfort in the medium term in patients who have undergone surgery for stress urinary incontinence by placing a suburethral sling. | 2 to 7 years after the surgery
  The primary endpoint of the research is the comparison of medians of the PPSSQ "discomfort and pain" score between women who underwent suburethral sling surgery and healthy female volunteers of the same age and menopausal status.

SECONDARY OUTCOMES:
To evaluate the quality of sexual life of patients who have undergone surgery for stress urinary incontinence using a suburethral sling. | 2 to 7 years after the surgery
  Comparison of medians of the PPSSQ "sexual health" score between women with suburethral sling surgery and healthy female volunteers.
Analyze the causes of discomfort and the characteristics of pain experienced by patients during intercourse. | 2 to 7 years after the surgery
  Analyse of PPSSQ answers to questions 5 and 6
To analyze the rate of non-sexually active patients after surgery, and the causes of this lack of sexuality. | 2 to 7 years after the surgery
  Analyse of PPSSQ answers to question 1
Compare sexual discomfort and quality of sexual life before/after suburethral sling surgery. | 2 to 7 years after the surgery
  Comparison of medians of the PPSSQ scores in the patient group before and after surgery

IPD SHARING:
Plan to Share IPD: No